CLINICAL TRIAL: NCT03188848
Title: A Randomized, Double-blind, Placebo Controlled, Dose Finding Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BPI-3016 in Healthy Subjects
Brief Title: Dose Escalating Study of BPI-3016 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTP-20211-01
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subject
MeSH Terms: interventions — BPI-3016

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPI-3016 (Experimental): Single-dose subcutaneous injection of BPI-3016 with escalating dose from 0.6 mg
  Interventions: Drug: BPI-3016
- Placebo (Placebo Comparator): Single-dose subcutaneous injection of placebo to match BPI-3016
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BPI-3016 — Single-dose subcutaneous injection of BPI-3016
  Arms: BPI-3016
Drug: Placebo — Single-dose subcutaneous injection of placebo to match BPI-3016
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose finding study evaluating the safety, pharmacokinetics and pharmacodynamics of subcutaneously injected BPI-3016 in Chinese healthy subjects.

DETAILED DESCRIPTION:
BPI-3016 is a novel analogue of glucagon-like peptide-1 (GLP-1) that developed for the treatment of type 2 diabetes mellitus. This is a randomized, double-blind, placebo-controlled, dose finding study evaluating the safety, pharmacokinetics and pharmacodynamics of subcutaneously injected BPI-3016 in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Subject's body mass index (BMI) is >=19 kilogram (kg)/meter(m)^2 and <=25 kg/m^2
* Male or female: if she is not pregnant (as confirmed by a test at screening and at other timepoints), not lactating, and at least one of the following conditions applies: a) cannot bear children OR b) agrees to follow contraception requirements defined in the protocol
* Capable of giving signed informed consent

Exclusion Criteria:

* Family history of multiple endocrine neoplasia, medullary carcinoma of the thyroid, or diabetes mellitus
* History of thymus disease, acute or chronic pancreatitis, or thyroid dysfunction
* History of gallstones, biliary motility dysfunction, cholecystitis or other gallbladder disease
* History of weight loss over 5% within 3 months of the study
* Abnormal blood pressure
* Abnormal blood routine, blood chemistry or test at screening
* Personal or family history of long QT syndrome, QT interval > 450 milliseconds (msec), or heart rate is >100 beats/min at Screening
* History of sensitivity or contraindication to any of the study medications or components thereof or a history of drug or other allergy
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result, or a positive test for Human immunodeficiency virus (HIV) antibody
* A positive pre-study drug/alcohol screen
* The subject participated in a clinical trial and received an investigational product within 90 days
* History of drug or other allergy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events and serious adverse events | 1 month
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement will be categorized as SAE
Plasma Concentrations of single-dose BPI-3016 | 15 days
  The concentration of BPI-3016 following single-dose administration was estimated
Tmax of single-dose BPI-3016 | 15 days
  Time of the maximum observed plasma concentration (tmax) following single-dose administration of BPI-3016 was estimated
AUC | 15 days
  The area under the concentration-time (AUC) curve from time zero to the last quantifiable concentration (0-last) and AUC (0-inf) of BPI-3016 were measured
T1/2 | 15 days
  The half-life (t1/2) of single-dose BPI-3016 was measured

SECONDARY OUTCOMES:
Change From Baseline in Fasting Plasma Glucose | 8 days
  Fasting Plasma Glucose was measured pre-dose at baseline, day 2, day 3, day 4, day 5, and day 8
Change From Baseline in 2 hours postprandial blood glucose | 8 days
  Fasting Plasma Glucose was measured pre-dose at baseline, day 2, day 3, day 4, day 5, and day 8

CONTACTS AND LOCATIONS:
Overall Officials: Kexin Li, Principal Investigator — Beijing Hospital; Lixin Guo, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No